CLINICAL TRIAL: NCT02450201
Title: A Pilot Study to Evaluate the Reproducibility of Magnetic Resonance (MR) Imaging With Hyperpolarized Pyruvate (13C) and Its Ability to Reflect Treatment Effects in Patients With Prostate Cancer
Brief Title: MRI With C13 Pilot Study Prostate Cancer
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Low accrual
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Rahul Aggarwal, Assistant Clinical Professor, University of California, San Francisco
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 125518
Record Dates: First submitted 2015-05-18; First posted 2015-05-21 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Pyruvic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Reproducibility (Experimental): Pyruvate injection followed by an MRI scan. 2-3 weeks after imaging #1: a second pyruvate injection followed by an MRI scan.
  Interventions: Drug: Pyruvate
- Part 2: Treatment Response (Experimental): Pyruvate injection followed by an MRI scan. 2 months after imaging #1: a second pyruvate injection followed by an MRI scan.
  Interventions: Drug: Pyruvate

INTERVENTIONS:
Drug: Pyruvate

SUMMARY:
This is a pilot clinical study of hyperpolarized pyruvate (13C) injection that includes the acquisition of magnetic resonance (MR) data and will be performed in men with localized prostate cancer. Part 1: Five patients will be evaluated for reproducibility of 13C HP MR imaging measurements obtained 2-3 weeks apart with no interim treatment. Part 2: Five patients will be evaluated for the change in 13C HP MR imaging measurements after 2 months of ADT.

13C HP MR data will be acquired in two parts of the study (which can occur simultaneously): Part 1: Patients will undergo imaging at baseline and will be repeated two to three weeks later (with no intervention in the interim) to evaluate reproducibility.

Part 2: Patients will undergo imaging at baseline, initiate androgen deprivation therapy, and undergo repeat imaging two months after initiation of ADT to evaluate the ability of the imaging to reflect a metabolic response to treatment.

The change in pyruvate/lactate ratio and lactate levels will be measured and compared to baseline at these timepoints.

ELIGIBILITY:
Inclusion Criteria:

* The subject has biopsy-proven adenocarcinoma of the prostate with intermediate to high risk disease by UCSF CAPRA scoring and possesses a Gleason 4 component to the tumor. Subjects will be enrolled either prior to radical prostatectomy (N=5) or prior to 2 months of androgen deprivation therapy (LHRH agonist +/- antiandrogen) followed by definitive radiation therapy as their primary treatment for prostate cancer (N=5).
* The subject is able and willing to comply with study procedures and provide signed and dated informed consent.
* At least 5 mm of tumor on biopsy (can have multiple cores to comprise 5 mm).
* The subject has concordant MRI/1H MRSI findings from a MR staging exam at UCSF performed prior to the 13C MRSI exam performed in this study with IMP, or is willing to undergo MRI/1H MRSI in connection with the study exam.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Laboratory criteria for protocol entry:
* Absolute neutrophil count (ANC) ≥1000 cells/µL
* Hemoglobin ≥9.0 gm/dL
* Platelets ≥75,000 cells/µL
* Estimated creatinine clearance ≥50 mL/min
* Total bilirubin ≤1.5x ULN (or if ≤4 gm/dL and direct bilirubin is WNL)
* Aspartate aminotransferase (AST) ≤1.5x ULN
* Alanine aminotransferase (ALT) ≤1.5x ULN
* Willing to use contraception during and for 1 month after completion of the study.
* For part 2 of the study: plans to initiate castrating therapy (with a GnRH antagonist, GnRH agonist, or orchiectomy). An antiandrogen may be started after initial imaging but can not be used prior to baseline imaging. An antiandrogen is allowed but not required.

Exclusion Criteria:

* The subject has received, or is scheduled to receive, another IMP from 1 month before to 1 month after inclusion in this study.
* Current or prior androgen deprivation therapy; previous use of a 5-α reductase inhibitor is allowed, provided it was discontinued at least one month prior to study entry.
* Poorly controlled hypertension, with blood pressure at study entry>160/100.
* Contraindication for or inability to tolerate MRI examination.
* Prostate biopsy within 12 weeks prior to study entry.
* BMI of less than 18.5 or greater than 32. Subject body weight should be less than or equal to 100 kg owing to limitations in the amount of IMP available.
* Congestive heart failure or New York Heart Association (NYHA) status≥2.
* A history of clinically significant EKG abnormalities, including QT prolongation, a family history of prolonged QT interval syndrome, or myocardial infarction (MI) less than 1 year ago with ensuing unstable EKG.
* Ongoing acute or chronic pulmonary bronchospastic disease, including a history of chronic obstructive pulmonary disease or asthma, with an exacerbation within the past year.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-10-12 (Actual); Primary Completion 2017-01-17 (Actual); Study Completion 2017-01-17 (Actual)

PRIMARY OUTCOMES:
Difference in peak lactate/pyruvate ratio | Baseline and 2-3 weeks after 1st image
Difference in peak lactate/pyruvate ratio | Baseline and 2 months after 1st image

SECONDARY OUTCOMES:
Pyruvate area under the curve (AUC) | Baseline and 2-3 weeks after 1st image
Lactate area under the curve (AUC) | Baseline and 2-3 weeks after 1st image
Pyruvate area under the curve (AUC) | Baseline and 2 months after 1st image
Lactate area under the curve (AUC) | Baseline and 2 months after 1st image
Safety As measured by Adverse Events | Up to 2 years
  As measured by Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Aggarwal, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States